CLINICAL TRIAL: NCT01014312
Title: Community-Based Depression Care Management for Elderly Primary Care Patients
Brief Title: Treatment for Depressed Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P30MH085943-02 (NIH); P30MH085943-02 (NIH); P30MH085943 (NIH); DATR A4-GPC (Other: National Institute of Mental Health)
Record Dates: First submitted 2009-11-03; First posted 2009-11-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depression Care Management (DCM) (Experimental): Participants will receive Depression Care Management.
  Interventions: Behavioral: Depression Care Management (DCM)
- Enhanced Care (Active Comparator): Participants will receive the standard of care from their primary care physicians enhanced by a summary of the study's diagnostic interview.
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Depression Care Management (DCM) — Depression Care Management (DCM) includes: 1. Monitoring the course of the depressive disorder; 2. Contacting the referring primary care physician (PCP) and offering information on the patients' current psychiatric status and medical complaints and the treatment recommended by published pharmacotherapy guidelines; 3. Determining the nature and extent of stressors affecting the patients' clinical status and functioning; 4. Psychoeducation concerning depression and depression treatment, working with the patient to select an appropriate treatment based on informed treatment preferences, and emphasizing treatment adherence; and 5. Supportive psychotherapy.
  Arms: Depression Care Management (DCM)
Behavioral: Enhanced Care — Primary Care Physicians will be informed by letter from a study psychologist of the participants' depression diagnosis and of suicidal ideation when present. They will have no direct assistance regarding depression treatment, but they will be educated on guideline-based antidepressant treatment recommendations. Moreover, research assistants will use a suicide risk protocol at baseline and at all follow-up assessment periods that mandates immediate contact with PCPs by telephone or beeper in cases with significant risk.
  Arms: Enhanced Care

SUMMARY:
This research study develop a collaborative depression care management model (C-DCM) that encourages collaboration between primary care physicians (PCPs) and trained social workers employed by community-based, public and nonprofit mental health clinics.

DETAILED DESCRIPTION:
Major depression affects 5%-9% of older primary care patients, is often chronic or recurrent and disabling, and leads to frequent use of medical services. Most depressed elders are treated by primary care physicians (PCPs) and prior research has shown that collaboration between primary care physicians and depression care managers is effective in treating depression. The challenge has been in securing third-party reimbursement for such services.

This research study will address this barrier by developing a collaborative depression care management model (C-DCM) that encourages collaboration between PCPs and trained social workers employed by community-based, public and nonprofit mental health clinics. In addition to developing C-DCM, a total of 112 primary care outpatients will participate in this study to test whether C-DCM is more effective than the standard of care in decreasing the severity of depression and disability experienced by older adults. Each subject will be randomized into either Usual Care or C-DCM. All subjects will be assessed at Baseline and at 2 and 4 months while the C-DCM subjects will also meet with social worker depression case managers bi-weekly over four months. If shown effective, C-DCM may bring to bear an available, yet untapped resource in the care of depressed elders.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older: This study focuses on the clinical complexities of late-life depression and its treatment. Family Services of Westchester (our partner community mental health agency) offers geriatric mental health counseling services to adults age 60 and older.
* Diagnosis of unipolar major depression
* MADRS score >=18: Depression of such severity in primary care patients requires treatment.
* CANE score >0: Reflects the presence of at least one unmet need in the domains of housing, self-care, safety, finances, benefits, legal matters, transportation, etc. and thus need for social services.
* Capacity to provide written consent for both research assessment and depression care management: PCPs will be asked to clinically evaluate prospective participants' capacity to consent and document it in their medical record.
* Working knowledge of English: Command in English sufficient for comprehending questionnaires of the study and/or for understanding the DCM therapists. English does not have to be the subject's first language.

Exclusion Criteria:

* Psychotic depression: This will be determined by the Structured Clinical Interview for DSM Disorders(SCID) assessment; presence of delusions and or hallucinations. This is a severe disorder typically referred for treatment to mental health specialists.
* Active suicidal ideation: This will be determined by the SCID and MADRS assessments. Older patients at these levels of risk for self-harm typically are referred to mental health specialists.
* Antisocial personality by Diagnostic and Statistical Manual of Mental Disorders (DSM)IV: This disorder will possibly interfere with adherence to research procedures and treatment.
* Significant Cognitive Impairment (MMSE score <24) or clinical diagnosis of dementia by DSM-IV: These conditions may limit the patient's ability to participate in treatment and require social service interventions exceeding those available through the proposed depression care management models.
* Current participation in specialist psychiatric care: Such patients will require the development of collaborative arrangements for depression care management which differ from those being tested in this study.
* Acute or severe medical illness: i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs often causing depression, e.g., steroids, reserpine, alpha-methyl-dopa, tamoxifen, vincristine.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Reduction in severity of depression over 16 weeks as measured by the Montgomery Asberg Depression Rating Scale (MADRS). | Measured at Baseline, 8 weeks, and 16 weeks

SECONDARY OUTCOMES:
Reduction in disability over 16 weeks as measured by the World Health Organization Disability Scale (WHODAS). | Measured at Baseline, 8 weeks, and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jo Anne Sirey, Ph.D., Principal Investigator — Weill Medical College of Cornell University; George S. Alexopoulos, M.D., Study Director — Weill Medical College of Cornell University
Locations (1):
- Westchester Medical Group Practices, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No